CLINICAL TRIAL: NCT05942625
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Studyto Evaluate the Safety, Tolerability and Pharmacokinetics of HS-10390 in Healthy Subjects
Brief Title: A First in Human Study to Evaluate Safety, Tolerability, Pharmacology of HS-10390 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10390-101
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: IgA Nephropathy; Focal Segmental Glomerulosclerosis
Keywords: HS-10390; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HS-10390 (Experimental): Single or multiple dosing of HS-10390 in a fastingstate
  Interventions: Drug: HS-10390 tablet
- Placebo (Experimental): Single or multiple dosing of placebo in a fastingstate
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: HS-10390 tablet — Oral administration of specified dose of HS-10390
  Arms: HS-10390
Drug: Placebo tablet — Oral administration of matching dose ofplacebo
  Arms: Placebo

SUMMARY:
The purpose of this first in human study is to evaluate the safety, tolerability, pharmacokinetics (PK),and pharmacodynamics (PD) of HS-10390 in healthy subjects.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single and multiple ascendingdose (SAD and MAD) study to evaluate the safety, tolerability, PK, and PD of different doses of HS-10390 tablet(s) in healthy subjects. During the SAD and MAD periods, there will be approximately 6and 3 sequential cohorts respectively. A sentinel dosing strategy will be used in the first cohort ofSAD. The MAD study will start after sufficient safety and PK data of SAD period are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of 18-45 years
* Have no reproductive potential; or agree to use a highly effective method ofcontraception, and refrain from donating sperm or eggs during the study period and forat least 6 months after last dosing
* Have signed the informed consent form approved by the IRB

Exclusion Criteria:

* History or evidence of clinically significant cardiovascular, pulmonary, endocrine,gastrointestinal, psychiatric, neurologic, hematological or metabolic diseases, especiallythose conditions that interfere with absorption, metabolism and/or excretion of the studydrug, determined by the investigator
* Have a clinically significant infection currently or within past 30 days, or have a history ofactive tuberculosis; or have positive screening test for infectious disease, includingtuberculosis, viral hepatitis, AIDS and syphilis
* Have a history of or current allergic disease
* Have a history of drug or alcohol abuse or currently positive test result(s) for alcohol ordrugs of abuse
* Smokers smoked ≥5 cigarettes per day within past 3 months or have a positive test resultfor nicotine
* Clinically significant abnormal physical examination, vital signs, clinical laboratory values,ECGs or imaging tests
* Pregnant or breastfeeding female subjects

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation | Day 1 up to Day 12 (SAD), Day 1 up to Day 28 (MAD)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
Time to reach Cmax (Tmax) | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
Half time (t½) | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
Apparent clearance (CL/F) | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
Apparent volume of distribution (Vz/F) | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
Accumulation ratio（Rac） | Day 14 up to Day 19 (MAD)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Affiliated to Southeast University, Nanjing, Jiangsu, China